CLINICAL TRIAL: NCT04820452
Title: A Multi-center, Randomized, Double-blind, Active-controlled Phase II Study to Evaluate the Efficacy and Safety of IBI302 in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Study of IBI302 in Patients With nAMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBI302A201
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — IBI302; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort 1 IBI302 treated with high dose level of IBI302 (Experimental): Drug: IBI302 4mg/eye;Intraocular injection
  Interventions: Biological: High dose IBI302
- Aflibercept (Active Comparator): Drug: Aflibercept 2mg/eye;Intraocular injection
  Interventions: Drug: Aflibercept
- cohort 1 IBI302 treated with low dose level of IBI302 (Experimental): Drug: IBI302 2mg/eye;Intraocular injection
  Interventions: Biological: Low dose IBI302

INTERVENTIONS:
Biological: Low dose IBI302 — Low dose IBI302 intravitreal injection given as every other month after three loading monthly injection
  Arms: cohort 1 IBI302 treated with low dose level of IBI302
Biological: High dose IBI302 — High dose IBI302 intravitreal injection given as every other month after three loading monthly injection
  Arms: cohort 1 IBI302 treated with high dose level of IBI302
Drug: Aflibercept — Intraocular injection
  Arms: Aflibercept

SUMMARY:
This is a multi-center, randomized, double-blind, active-controlled study to evaluate the efficacy and safety of IBI302 in subjects with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion criteria

1. Male or female patient ≥ 50 yrs. of age.
2. Active subfoveal or parafoveal CNV secondary to neovascular AMD.
3. BCVA score of 24-73 letters using ETDRS charts in the study eye.
4. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.

Exclusion criteria

1. Concomitant diseases that may cause subjects fail to respond to the treatment or confuse the interpretation of the study results;
2. Presence of uncontrolled glaucoma in the study eye (defined as IOP≥25mmHg despite the standardized treatment);
3. Presence of active intraocular or periocular inflammation or infection;
4. Prior any treatment of following in the study eye:

   1. Anti-VEGF therapy or anti-complement therapy within 3 months prior to screening;
   2. Laser photocoagulation within 3 months prior to screening;
   3. Photodynamic therapy or vitreoretinal surgery;
   4. Intraocular glucocorticoid injection within 6 months prior to enrollment;
5. Presence of any systemic disease: including but not limited toactive infections (such as active viral hepatitis); unstable angina; cerebrovascular accident or transient cerebral ischemia (within 6 months prior to selection); myocardial infarction (within 6 months prior to selection); serious arrhythmia requiring medical treatment; liver, kidney or metabolic diseases; or malignant tumor;
6. History of severe hypersensitivity/allergy to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
7. Pregnant or lactating women or women preparing to become pregnant or breastfeeding during the study period;
8. Participated in any clinical study of any other drug within three months prior to enrollment, or attempted to participate in other drug trials during the study;
9. Other conditions unsuitable for enrollment judged by investigators

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
The visual efficacy of IBI302 | Baseline to week 36

SECONDARY OUTCOMES:
other visual effects of IBI302 | Baseline to week 52
  the proportion if BCVA improvement ≥0,5,10 or 15 letters at week 12, 28, 36 and 52.
the anatomical effects of IBI302 on OCT | Baseline to week 52
  the mean change of central subfield thickness from BL to week 52 at week 12, 28, 36 and 52
the anatomical effects of IBI302 on FFA | Baseline to week 52
  the change of CNV area, CNV leakage area, total lesion area from BL to week 36 or 52
the safety of IBI302 | Baseline to week 52
  the incidence of ocular AE or any systemic AE, TEAE, SAE
Immunogenicity of IBI302 | Baseline to week 52
  the positive rate of anti-drug antibody and neutralizing antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Innovent Biologics (Suzhou) Co,Ltd., Suzhou, Jiangsu, China